CLINICAL TRIAL: NCT07337564
Title: A Clinical Study Evaluating the Efficacy and Safety of SHR-1139 Injection in Adult Patients With Ulcerative Pyoderma Gangrenosum
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong First Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-IIT-SHR1139
Record Dates: First submitted 2025-12-17; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pyoderma Gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1139 injection group (Experimental)
  Interventions: Drug: SHR-1139 Injection

INTERVENTIONS:
Drug: SHR-1139 Injection — SHR-1139 Injection

SUMMARY:
This study was designed to assess the therapeutic efficacy and safety of SHR-1139 Injection in adult patients with ulcerative pyoderma gangrenosum.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 years old at the time of signing the informed consent form (ICF).
* Diagnosed with ulcerative PG during screening, and requiring systemic treatment as assessed by the investigator.
* At screening and baseline, there is at least one measurable PG ulcer. If a subject has more than one PG ulcer, the investigator will select the target PG ulcer.
* Subjects voluntarily sign informed consent form (ICF) prior to the commencement of any procedures related to the study, are able to communicate smoothly with the investigator, understand and are willing to complete the study in strict compliance with the requirements of this clinical study protocol.
* Adequate organ and bone marrow function.
* Female subjects of childbearing potential or male subjects whose partners are females of childbearing potential shall have no plans for childbearing, sperm/egg donation from the time of signing the informed consent form until 72 weeks after the last dose, and shall voluntarily adopt effective contraceptive measures (including their partners). Female subjects must have a negative pregnancy test result during the screening period and before randomization and drug administration, and must not be breastfeeding.

Exclusion Criteria:

* At screening, the clinical manifestations are other ulcers or other similar skin lesions caused by non-PG diseases;
* There is a significant medical history or underlying disease that affects safety.
* A history of allergy to the study drug or any component of the study drug before screening.
* A history of alcohol abuse or illegal drug abuse within one year before screening;
* Having donated approximately 500 mL of blood within 8 weeks before baseline or having plans to donate blood during the study.
* Other circumstances that the investigator judges may affect the evaluation of the safety and efficacy of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects whose target PG ulcer achieves complete closure (100% reduction in PG area, PGAR-100) at Week 12. | Week 12

SECONDARY OUTCOMES:
The proportion of subjects whose target PG ulcer achieves 50% closure (50% reduction in PG area, PGAR-50) at Week 12 | Week 12
The proportion of subjects whose target PG ulcer achieves complete closure (100% reduction in PG area, PGAR-100) at any time point before Week 26; | up to Week 26
adverse events(AEs) | up to Week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Hospital Affiliated to Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No